CLINICAL TRIAL: NCT02027311
Title: Etomidate With Meperidine vs Midazolam With Meperidine for Sedation During Endodscopic Retrograde Cholangiopancreatogram (ERCP)
Brief Title: Etomidate vs. Midazolam for Sedation During ERCP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cheju Halla General Hospital (Other)
Responsible Party: Principal Investigator, Byung Hyo Cha, MD, Director of Endoscopy clinic, Digestive Disease Center, Department of Internal Medicine, Cheju Halla General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ETOMI-1
Record Dates: First submitted 2013-04-16; First posted 2014-01-06 (Estimated); Results first posted 2015-06-29 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Choledocholithiasis; Cholangiocarcinoma; Pancreatitis; Pancreatic Cancer
Keywords: Endoscopic Retrograde Cholangiopancreatography (ERCP); Conscious Sedation; etomidate; midazolam
MeSH Terms: conditions — Choledocholithiasis; Cholangiocarcinoma; Pancreatitis; Pancreatic Neoplasms | interventions — Etomidate; Midazolam; Meperidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Etomidate (Experimental): This cohort would be administered etomidate with meperidine. The initial dose of etomidate is 0.1mg/kg IV and meperidine, 25mg. Additional dose of etomidate is 2mg(1cc). In old age cased, more than 65 years old, 30% of initial dose discounted.
  Interventions: Drug: Etomidate; Drug: Meperidine
- Midazolam (Experimental): This cohort would be administered midazolam with meperidine. The initial dose of midazolam is 0.06mg/kg IV and meperidine 50mg IV. Additional dose is 1mg of midazolam. In the elders, more than 65 years old, initial dose was declined to 70%.
  Interventions: Drug: Midazolam; Drug: Meperidine

INTERVENTIONS:
Drug: Etomidate — This cohort would be administered etomidate with meperidine. The initial dose of etomidate is 0.1mg/kg IV and meperidine, 25mg. Additional dose of etomidate is 2mg(1cc). In old age cased, more than 65 years old, 30% of initial dose discounted.
  Other Names: Etomidate lipro IV
  Arms: Etomidate
Drug: Midazolam — This cohort would be administered midazolam with meperidine. The initial dose of midazolam is 0.06mg/kg IV and meperidine 50mg IV. Additional dose is 1mg of midazolam. In the elders, more than 65 years old, initial dose was declined to 70%.
  Arms: Midazolam
Drug: Meperidine — Both groups were administered same dose of meperidinie 50mg. Then elders > 80 years old were administered 25mg iv bolus.
  Other Names: Pethidine

SUMMARY:
Recently up-coming drug, etomidate which is a modulator of GABA(gamma-Aminobutyric acid)-A receptor has been known that it maintains the appropriate sedative levels and affects little effects on respiratory system.

The investigators are now trying to investigate that etomidate with meperidine combination regimen is superior to the midazolam with meperidine more effective and less harm on sedation during the ERCP procedure.

DETAILED DESCRIPTION:
ERCP (Endoscopic retrograde cholangiopancreatogram) is an uncomfortable and time-consuming procedure compared to other endoscopic procedures. Most ERCP procedure had been performed in sedation using tranquilizers and pain-killers.

Until recently, midazolam and opioid combination regimen recognized as a standard therapy is widely used, but the sedative effect is insufficient and intermittent paradoxical reaction has been questioned. Another drug, such as propofol, has been known that the sedative effect is superior one of the midazolam but disappointed due to narrow therapeutic range of respiratory distress and absence of antagonist. Meanwhile, recently up-coming drug, etomidate which is a modulator of GABA-A receptor has been known that it maintains the appropriate sedative levels and affects little effects on respiratory system.

For these advantages, this short acting sedative drug has been widely used in the emergency room during minor operation and in the operation room for induction. However, research on the efficacy during ERCP was not yet published.

In this regards, the purpose of the investigators study is to prove the efficacy of etomidate for sedation and to establish new evidence based sedation guidelines during ERCP procedure.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are scheduled diagnositic or therapeutic ERCP.
* Age : more than 20 and less than 90 years old
* ASA(American Society of Anesthesiologists) classificiation : I, II, III

Exclusion Criteria:Patients following

* Refuse to be enrolled
* ASA American Society of Anesthesiologists)classification IV, V
* Breast feeder
* The mentally ill
* Drug abuser
* Hypersensitivity to sedative or opioids
* Alcohol intoxication or dependency
* Body mass index (BMI) 36kg/m2 or more
* Unstable vital sign

  1. tachypnea, respiration rate more than 25/min or less than 10/min
  2. Oxygen saturation : 90% or less
  3. Systolic blood pressure : less than 90 mmHg or more than 180 mmHg
  4. Diastolic blood pressure : less than 50 mmHg or more than 100 mmHg
  5. Heart rate : more than 120 beat/min or less than 50 beat/min.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: BYUNG HYO CHA, Dr., Study Chair — Cheju Halla General Hospital, Doreongno 65, Jeju-si Jeju Special Self-Governing Province, Korea 690-766
Locations (1):
- 1Digestive Disease Center and Department of Internal Medicine, Cheju Halla General Hospital, Jeju City, Jeju Special Self-Governing Province, South Korea

REFERENCES:
- [Background] Standards of Practice Committee of the American Society for Gastrointestinal Endoscopy; Lichtenstein DR, Jagannath S, Baron TH, Anderson MA, Banerjee S, Dominitz JA, Fanelli RD, Gan SI, Harrison ME, Ikenberry SO, Shen B, Stewart L, Khan K, Vargo JJ. Sedation and anesthesia in GI endoscopy. Gastrointest Endosc. 2008 Nov;68(5):815-26. doi: 10.1016/j.gie.2008.09.029. No abstract available. PMID 18984096
- [Background] Yamazaki N, Ogawa K. [Dopamine-beta-hydroxylase (DBH)]. Kokyu To Junkan. 1976 Nov;24(11):949-55. No abstract available. Japanese. PMID 1034320
- [Background] Bell GD. Review article: premedication and intravenous sedation for upper gastrointestinal endoscopy. Aliment Pharmacol Ther. 1990 Apr;4(2):103-22. doi: 10.1111/j.1365-2036.1990.tb00455.x. PMID 2104078
- [Background] Galletly D, Forrest P, Purdie G. Comparison of the recovery characteristics of diazepam and midazolam. Br J Anaesth. 1988 Apr;60(5):520-4. doi: 10.1093/bja/60.5.520. PMID 3377928
- [Background] Yuksel O, Parlak E, Koklu S, Ertugrul I, Tunc B, Sahin B. Conscious sedation during endoscopic retrograde cholangiopancreatography: midazolam or midazolam plus meperidine? Eur J Gastroenterol Hepatol. 2007 Nov;19(11):1002-6. doi: 10.1097/MEG.0b013e3282cf5167. PMID 18049171
- [Background] Radaelli F, Meucci G, Terruzzi V, Spinzi G, Imperiali G, Strocchi E, Lenoci N, Terreni N, Mandelli G, Minoli G. Single bolus of midazolam versus bolus midazolam plus meperidine for colonoscopy: a prospective, randomized, double-blind trial. Gastrointest Endosc. 2003 Mar;57(3):329-35. doi: 10.1067/mge.2003.104. PMID 12612511
- [Background] Reimann FM, Samson U, Derad I, Fuchs M, Schiefer B, Stange EF. Synergistic sedation with low-dose midazolam and propofol for colonoscopies. Endoscopy. 2000 Mar;32(3):239-44. doi: 10.1055/s-2000-134. PMID 10718390
- [Background] Sipe BW, Rex DK, Latinovich D, Overley C, Kinser K, Bratcher L, Kareken D. Propofol versus midazolam/meperidine for outpatient colonoscopy: administration by nurses supervised by endoscopists. Gastrointest Endosc. 2002 Jun;55(7):815-25. doi: 10.1067/mge.2002.124636. PMID 12024134
- [Background] Riker RR, Shehabi Y, Bokesch PM, Ceraso D, Wisemandle W, Koura F, Whitten P, Margolis BD, Byrne DW, Ely EW, Rocha MG; SEDCOM (Safety and Efficacy of Dexmedetomidine Compared With Midazolam) Study Group. Dexmedetomidine vs midazolam for sedation of critically ill patients: a randomized trial. JAMA. 2009 Feb 4;301(5):489-99. doi: 10.1001/jama.2009.56. Epub 2009 Feb 2. PMID 19188334
- [Background] Jung M, Hofmann C, Kiesslich R, Brackertz A. Improved sedation in diagnostic and therapeutic ERCP: propofol is an alternative to midazolam. Endoscopy. 2000 Mar;32(3):233-8. doi: 10.1055/s-2000-96. PMID 10718389
- [Background] Falk J, Zed PJ. Etomidate for procedural sedation in the emergency department. Ann Pharmacother. 2004 Jul-Aug;38(7-8):1272-7. doi: 10.1345/aph.1E008. Epub 2004 Jun 1. PMID 15173551
- [Background] Hunt GS, Spencer MT, Hays DP. Etomidate and midazolam for procedural sedation: prospective, randomized trial. Am J Emerg Med. 2005 May;23(3):299-303. doi: 10.1016/j.ajem.2005.02.042. PMID 15915401
- [Background] Denny MA, Manson R, Della-Giustina D. Propofol and Etomidate are Safe for Deep Sedation in the Emergency Department. West J Emerg Med. 2011 Nov;12(4):399-403. doi: 10.5811/westjem.2011.5.2099. PMID 22224127
- [Background] Miner JR, Martel ML, Meyer M, Reardon R, Biros MH. Procedural sedation of critically ill patients in the emergency department. Acad Emerg Med. 2005 Feb;12(2):124-8. doi: 10.1197/j.aem.2004.08.054. PMID 15692132
- [Background] Ruth WJ, Burton JH, Bock AJ. Intravenous etomidate for procedural sedation in emergency department patients. Acad Emerg Med. 2001 Jan;8(1):13-8. doi: 10.1111/j.1553-2712.2001.tb00539.x. PMID 11136141
- [Background] Mandt MJ, Roback MG, Bajaj L, Galinkin JL, Gao D, Wathen JE. Etomidate for short pediatric procedures in the emergency department. Pediatr Emerg Care. 2012 Sep;28(9):898-904. doi: 10.1097/PEC.0b013e318267c768. PMID 22929142
- [Background] Terui T, Inomata M. Administration of additional analgesics can decrease the incidence of paradoxical reactions in patients under benzodiazepine-induced sedation during endoscopic transpapillary procedures: prospective randomized controlled trial. Dig Endosc. 2013 Jan;25(1):53-9. doi: 10.1111/j.1443-1661.2012.01325.x. Epub 2012 Jun 11. PMID 23286257
- [Background] Honan VJ. Paradoxical reaction to midazolam and control with flumazenil. Gastrointest Endosc. 1994 Jan-Feb;40(1):86-8. doi: 10.1016/s0016-5107(94)70020-6. No abstract available. PMID 8163147
- [Background] Ladas SD, Aabakken L, Rey JF, Nowak A, Zakaria S, Adamonis K, Amrani N, Bergman JJ, Boix Valverde J, Boyacioglu S, Cremers I, Crowe J, Deprez P, Dite P, Eisen M, Eliakim R, Fedorov ED, Galkova Z, Gyokeres T, Heuss LT, Husic-Selimovic A, Khediri F, Kuznetsov K, Marek T, Munoz-Navas M, Napoleon B, Niemela S, Pascu O, Perisic N, Pulanic R, Ricci E, Schreiber F, Svendsen LB, Sweidan W, Sylvan A, Teague R, Tryfonos M, Urbain D, Weber J, Zavoral M; European Society of Gastrointestinal Endoscopy Survey of National Endoscopy Society Members. Use of sedation for routine diagnostic upper gastrointestinal endoscopy: a European Society of Gastrointestinal Endoscopy Survey of National Endoscopy Society Members. Digestion. 2006;74(2):69-77. doi: 10.1159/000097466. Epub 2006 Nov 27. PMID 17135728
- [Background] Cohen LB, Wecsler JS, Gaetano JN, Benson AA, Miller KM, Durkalski V, Aisenberg J. Endoscopic sedation in the United States: results from a nationwide survey. Am J Gastroenterol. 2006 May;101(5):967-74. doi: 10.1111/j.1572-0241.2006.00500.x. PMID 16573781
- [Background] Riphaus A, Rabofski M, Wehrmann T. Endoscopic sedation and monitoring practice in Germany: results from the first nationwide survey. Z Gastroenterol. 2010 Mar;48(3):392-7. doi: 10.1055/s-0028-1109765. Epub 2010 Feb 5. PMID 20140841
- [Background] Fanti L, Agostoni M, Casati A, Guslandi M, Giollo P, Torri G, Testoni PA. Target-controlled propofol infusion during monitored anesthesia in patients undergoing ERCP. Gastrointest Endosc. 2004 Sep;60(3):361-6. doi: 10.1016/s0016-5107(04)01713-4. PMID 15332024
- [Background] Chen WX, Lin HJ, Zhang WF, Gu Q, Zhong XQ, Yu CH, Li YM, Gu ZY. Sedation and safety of propofol for therapeutic endoscopic retrograde cholangiopancreatography. Hepatobiliary Pancreat Dis Int. 2005 Aug;4(3):437-40. PMID 16109532
- [Background] Kongkam P, Rerknimitr R, Punyathavorn S, Sitthi-Amorn C, Ponauthai Y, Prempracha N, Kullavanijaya P. Propofol infusion versus intermittent meperidine and midazolam injection for conscious sedation in ERCP. J Gastrointestin Liver Dis. 2008 Sep;17(3):291-7. PMID 18836622
- [Background] Carrasco G. Instruments for monitoring intensive care unit sedation. Crit Care. 2000;4(4):217-25. doi: 10.1186/cc697. Epub 2000 Jul 13. PMID 11094504
- [Background] Frade Mera MJ, Guirao Moya A, Esteban Sanchez ME, Rivera Alvarez J, Cruz Ramos AM, Bretones Chorro B, Vinas Sanchez S, Jacue Izquierdo S, Montane Lopez M. [Analysis of 4 sedation rating scales in the critical patient]. Enferm Intensiva. 2009 Jul-Sep;20(3):88-94. doi: 10.1016/s1130-2399(09)72588-x. Spanish. PMID 19775565

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligibility was evaluated for all patients with a scheduled ERCP procedure in the Cheju Halla General Hospital during the study period from May 15 2013 to Aug 19 2013. Sample size estimated 26 of each groups for reject null hypothesis with probability (power) 0.8 and Type I error is 0.05.
Pre-assignment Details: 68 patients were enrolled and 35 were assigned in the MDZ group and 33 were in the ETM group. In ETM group, 1 case was dropped due to hypotension and 2 were desaturation. And 1 cases was dropped due to tachycardia and 1 were desaturation in MDZ group.
Period: Overall Study
Arm/Group | Etomidate | Midazolam
Started | 33 | 35
Completed | 30 (1 case was dropped due to hypotension and 2 were desaturation.) | 33 (1 cases was dropped due to tachycardia and 1 were desaturation.)
Not Completed | 3 | 2
Not completed — Protocol Violation | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Etomidate | Midazolam | Total
Number analyzed (Participants) | 30 | 33 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (15.7) | 71.6 (11.5) | 70.9 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 35
  Male | 14 | 14 | 28
Body Mass Index (kg/square of m.) [Mean (Standard Deviation); unit: kg/square of m.] | 23.7 (3.5) | 22.6 (4.31) | 23.1 (3.9)
Procedure Time (min) [Mean (Standard Deviation); unit: min] | 27.6 (14.9) | 32.8 (13.4) | 30.4 (14.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Intervention
Description: The frequency of intervention which was defined as any restraint of the patient's head, arms, or legs if they became agitated, or if patient movement was not controlled with verbal instruction from the endoscopist during the whole intraoperative phases.
Time Frame: Throughout the whole ERCP procedure
Measure: Mean (Standard Deviation); unit: Number of intervention
Arm/Group | Etomidate | Midazolam
Number analyzed (Participants) | 30 | 33
Number of intervention | 1.9 (3.1) | 7.5 (6.8)
Statistical Analysis 1: Comparison: Etomidate vs Midazolam; If the true difference in the experimental and control means is 4, total 26 experimental subjects and 26 control subjects was required to reject the null hypothesis that the means of the primary outcome values of experimental and control groups are equal with probability (power) 0.8. The Type I error probability associated with this test of this null hypothesis is 0.05; Test type: Superiority or Other; p = 0.05, Regression, Logistic — For two-sided tests, p < 0.05 was considered statistically significant; Logistic regression model used to identify the factors related to the presence of intervention (frequency of intervention = 0, vs. ≥ 1)

2. Secondary Outcome: Event of Hypoxia
Description: Hypoxia defined as peripheral blood oxygen saturation measured by pulse oxymeter < 90%
Time Frame: Every 5min in Preoperative, intraoperative phase and 15 min in Recovery phase
Measure: Number; unit: Hypoxia events
Arm/Group | Midazolam | Etomidate
Number analyzed (Participants) | 33 | 30
Hypoxia events | 19 | 27
Statistical Analysis 1: Comparison: Midazolam vs Etomidate; All the continuous variables were compared using the Mann-Whitney U test and dichotomous categorical variables was used and the Pearson chi-square with Fisher exact test. We used the linear mixed model to compare the differences of paired data, such as mean values of RR, SpO2, MAP, HR, and RSS at different time points of the two different sedation groups. For two-sided tests, p < 0.05 was considered statistically significant; Test type: Superiority or Other; p = 0.002, Regression, Logistic — Logistic regression model were used in univariate and corrected multivariate analyses to identify the factors related to the primary outcome variables, such as, presence of intervention (frequency of intervention = 0, vs. ≥ 1); Odds Ratio (OR) = 11.09, 95% CI 2-sided [2.41 to 50.94]

ADVERSE EVENTS:
Time Frame: BP, RR, HR, and SpO2 were monitored at 5-minute intervals after the baseline measurements until the termination of the ERCP. The baseline measurements were obtained at least 15 minutes before any medication was administered to patients.
Description: Additional probable side events, such as, paradoxic reaction in MDZ group, and myoclonus in ETM group were counted during the whole 3 phases of procedure.
Arm/Group | Etomidate | Midazolam
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/33
Other Adverse Events (participants affected / at risk) | 0/30 | 0/33

LIMITATIONS AND CAVEATS:
1. To standardize proper sedation level we used Ramsay Sedation Scale but this scale could be calculated subjectively.
2. Double blindness was not applied strictly because of quite different pharmacodynamics of two experimental drugs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No